CLINICAL TRIAL: NCT01213823
Title: Risk Of Severe Hepatic Injury In Patients With Invasive Candidiasis Treated With Echinocandins
Status: Terminated | Type: Observational
Why Stopped: The study was terminated on May 5, 2011, due to methodological issues. The decision to terminate the study was not based on any safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8851024
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Invasive Candidiasis; Candidemia
Keywords: invasive candidiasis; candidemia; severe hepatic injury; echinocandins; anidulafungin; caspofungin; micafungin
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Potential cases were defined as patients with a diagnosis of severe hepatic injury identified in the acute-care inpatient cohort using ICD-9 codes associated with the case definition of severe liver injury. Case status was validated by a Consultant Gastroenterologist blinded to study drug exposure via medical record review using an apriori algorithm. Only validated cases were included in the analysis (N=69)
  Interventions: Other: Does not apply
- Controls: Controls were defined as patients without a diagnosis of severe hepatic injury (i.e. with no ICD-9 codes associated with the case definition of severe liver injury) selected at random from the same acute-care inpatient cohort as cases (N=467)
  Interventions: Other: Does not apply

INTERVENTIONS:
Other: Does not apply — This is a non-interventional study, therefore the intervention type / name do not apply
  Groups: Cases
Other: Does not apply — This is a non-interventional study, therefore the intervention type / name do not apply
  Groups: Controls

SUMMARY:
The purpose of this study is to estimate the relative risk of severe hepatic injury in hospitalized patients with invasive candidiasis and candidemia who received anidulafungin, compared to patients who received caspofungin and/or micafungin.

ELIGIBILITY:
Inclusion Criteria:

* Acute-care inpatients;
* Aged 18 years or older;
* At least one dose of echinocandin therapy during the hospitalization;
* Primary or secondary ICD-9 discharge diagnosis of invasive candidiasis / candidemia.

Exclusion Criteria:

* < 18 years of age;
* No recorded echinocandin therapy during hospitalization;
* Acetaminophen hepatotoxicity;
* Pre-existing autoimmune hepatitis;
* Autoimmune/metabolic liver disease;
* Primary biliary cirrhosis;
* Primary sclerosing cholangitis and orthotopic liver transplantation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute-care inpatients aged 18 years or older, with at least one dose of echinocandin antifungal therapy during the hospitalization and a primary or secondary ICD-9 discharge diagnosis of invasive candidiasis / candidemia identified in the Premier's PerspectiveTM Comparative Database (PCD) from 01 June 2006 to 30 June 2008.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851024&StudyName=Risk%20Of%20Severe%20Hepatic%20Injury%20In%20Patients%20With%20Invasive%20Candidiasis%20Treated%20With%20Echinocandins

RESULTS

PARTICIPANT FLOW:
Groups:
- Cases: Potential cases were to be defined as participants with invasive candidiasis (candidiasis of the lung, disseminated candidiasis, candidal endocarditis, candidal meningitis, candidal enteritis, or candidiasis of unspecified site) with severe hepatic injury (acute/subacute necrosis of liver, hepatic coma, hepatorenal syndrome, or hepatitis unspecified) classified into one of the following categories: 1) acute liver failure (associated with encephalopathy and/or coagulopathy in absence of underlying liver disease); 2) Hy's Law Criteria (serum alanine transaminase [ALT] levels greater than [>]3 times the upper limit of normal [xULN] and total bilirubin >2 xULN, with absence of alkaline phosphatase elevation; 3) serum ALT levels greater than or equal to (≥)10 xULN; 4) ALT levels >3 xULN and less than (<)10 xULN; or 5) as determined by clinician.
- Controls: Controls were to be defined as participants with invasive candidiasis (candidiasis of the lung, disseminated candidiasis, candidal endocarditis, candidal meningitis, candidal enteritis, or candidiasis of unspecified site) without a diagnosis of severe hepatic injury.
Period: Overall Study
Arm/Group | Cases | Controls
Started | 69 | 467
Completed | 69 | 467
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 69 | 467 | 536
Age, Customized [Number; unit: Participants]
  18-24 years | 1 | 12 | 13
  25-34 years | 1 | 26 | 27
  35-44 years | 5 | 42 | 47
  45-54 years | 15 | 73 | 88
  55-64 years | 16 | 76 | 92
  65-74 years | 18 | 111 | 129
  Greater than or equal to (>=) 75 years | 13 | 127 | 140
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 245 | 274
  Male | 40 | 222 | 262

OUTCOME MEASURES:

1. Primary Outcome: Number of Any Severe Hepatic Injury Cases and Matched Controls
Description: Severe hepatic injury (acute/subacute necrosis of liver, hepatic coma, hepatorenal syndrome, or hepatitis unspecified) classified as: 1) acute liver failure (associated with encephalopathy and/or coagulopathy in absence of underlying liver disease); 2) Hy's Law Criteria (serum alanine transaminase [ALT] levels greater than [>]3 times the upper limit of normal [ULN] and direct bilirubin >2 times ULN and absence of alkaline phosphatase elevation); 3) ALT levels greater than or equal to (≥) 10 times ULN; 4) ALT levels >3 times ULN and less than (<) 10 times ULN; or 5) classified by clinician. Disease Related Group (DRG) severity of illness coding was reported for severe hepatic injury cases and matched controls.
Time Frame: 01 June 2006 to 30 June 2008 (up to 25 Months)
Population: Acute-care participants, with at least 1 dose of echinocandin antifungal therapy and a primary or secondary International Classification of Diseases 9 (ICD-9).
Measure: Number; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 69 | 467
Participants
  DRG Severity Coding 1 | 0 | 1
  DRG Severity Coding 2 | 0 | 10
  DRG Severity Coding 3 | 1 | 66
  DRG Severity Coding 4 | 68 | 389

ADVERSE EVENTS:
Description: In this retrospective observational study, adverse events were not collected as a part of this study.
Arm/Group | Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study results were invalidated due to lack of temporality, a critical methodological element of the study that was never established for the majority of the cases of severe hepatic injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.